CLINICAL TRIAL: NCT07021625
Title: Use of CBT-I Based Chatbot for Assisted Treatment in Patients With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N202306054
Record Dates: First submitted 2025-06-03; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Insomnia; Depression/Anxiety
Keywords: Insomnia; Chatbot; CBT; Cognitive behavioral therapy; Cognitive behavioral therapy for insomnia; CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The experimental group will receive four weeks of cognitive behavioral therapy for insomnia via a chatbot, while the control group will be treated as usual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): four weeks of cognitive behavioral therapy for insomnia via a chatbot
  Interventions: Device: Kunbot
- Control group (Placebo Comparator): treated as usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Device: Kunbot — A chatbot designed based on cognitive behavioral therapy for insomnia
  Arms: Experimental group
Other: Treatment as usual — Treatment as usual
  Arms: Control group

SUMMARY:
The recent lifestyle has put many people in a state of high stress, and the outbreak of COVID-19 in recent years has caused a steady increase in the number of people diagnosed with "Coronasomnia" (Covid-somnia) after recovering from the disease. For reasons outlined above, a lot number of people were suffering from Insomnia. To propose some method to improve patients' sleep disorders become a popular research issue. The American Academy of Sleep Medicine strongly recommends using the Cognitive Behavioral Therapy for insomnia (CBT-I) method, one of the non-pharmacological treatments for insomnia. However, CBT-I is primarily a physical therapy, so patients may not be able to access this therapy due to time and location constraints. This project aims to combine the technology of Cognitive Behavioral Therapy for Insomnia (CBT-I) and chatbot to help insomnia patients learn more about their sleep habits and improve their sleep quality at home through remote access. Investigators will design a friendly chatbot based on the CBT-I concept to assist insomnia patients to improve their sleep quality and life quality.

This project will be executed at Taipei Municipal Wanfang Hospital. Patients of insomnia will be referred by the attending physician from outpatient clinic. It is estimated that 120 patients will be enrolled, 60 in the experimental group and 60 in the control group. The experimental group will receive four weeks of cognitive behavioral therapy for insomnia via a chatbot, while the control group will be treated as usual. Patients will be assessed for improvement in sleep severity at the end of four weeks and follow up after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Significant insomnia symptoms, including difficulty initiating sleep, difficulty maintaining sleep, early-morning awakening.

   The sleep difficulty occurs at least three nights per week and is present for at least 3 months.
3. Patient possess a personal internet-connected cell phone or communicator.

Exclusion Criteria:

1. Unwilling to participate in this research.
2. Have poor cognitive function and cannot understand the content of the questionnaire; or cannot complete the test due to their physical condition
3. Comorbid with schizophrenia, bipolar disorder, or substance use disorder
4. Medications received have been adjusted in the past one month or will be adjusted during experiment
5. Those who received in the past one month or will receive during experiment treatments such as: psychotherapy, cranial electrical stimulation, repetitive transcranial magnetic stimulation, transcranial direct current stimulation, or nutraceuticals aimed at improving mood or insomnia.
6. Suicidal patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index | From enrollment to the end of treatment at 4 weeks
  Value: 0~21, higher score means a worse outcome

SECONDARY OUTCOMES:
Patient Health Questionnaire | From enrollment to the end of treatment at 4 weeks
  Value: 0~27, higher score means a worse outcome
Beck Depression Inventory | From enrollment to the end of treatment at 4 weeks
  Value: 0~63, higher score means a worse outcome
Beck Anxiety Inventory | From enrollment to the end of treatment at 4 weeks
  Value: 0~63, higher score means a worse outcome
Brief Symptom Rating Scale | From enrollment to the end of treatment at 4 weeks
  Value: 0~20, higher score means a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- WanFang Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
This project aims to combine the technology of Cognitive Behavioral Therapy for Insomnia (CBT-I) and chatbot to help insomnia patients learn more about their sleep habits and improve their sleep quality at home through remote access. We will design a friendly chatbot based on the CBT-I concept to assist insomnia patients to improve their sleep quality and life quality.
  Patients of insomnia will be referred by the attending physician from outpatient clinic. It is estimated that 120 patients will be enrolled, 60 in the experimental group and 60 in the control group. The experimental group will receive four weeks of cognitive behavioral therapy for insomnia via a chatbot, while the control group will be treated as usual. Patients will be assessed for improvement in sleep severity at the end of four weeks and follow up after 12 weeks.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: July 2023-December 2025